CLINICAL TRIAL: NCT01256957
Title: Assessing the Impact of Wood Stove Interventions on Air Quality
Brief Title: Effect of HEPA Air Filters on Subclinical Markers of Cardiovascular Health
Acronym: WEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: University of British Columbia (Other); Health Canada (Other Government); Ministry of Environment, British Columbia (Other)
Responsible Party: Principal Investigator, Ryan Allen, Associate Professor, Simon Fraser University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 869329
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2010-12

CONDITIONS: Endothelial Function; Oxidative Stress; Systemic Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indoor air HEPA filtration (Active Comparator): HEPA filters operating in the participant's bedroom and living room.
  Interventions: Device: HEPA filter
- Control (No Intervention): Control

INTERVENTIONS:
Device: HEPA filter
  Other Names: Honeywell model 50300; Honeywell model 18150
  Arms: Indoor air HEPA filtration

SUMMARY:
The purpose of this study is to evaluate the ability of portable high efficiency particle air (HEPA) filters to reduce exposures to PM2.5 and woodsmoke air pollution indoors and to improve subclinical indicators of microvascular function, systemic inflammation, and oxidative stress among healthy adult participants.

DETAILED DESCRIPTION:
The investigators will use portable HEPA filters in a single-blind randomized crossover design. Each participant's home will be monitored for two consecutive seven-day periods, during which time two HEPA units (one in the bedroom and one in the main living room) will be operated indoors. During one 7-day period the HEPA filters will be operated normally, and during the other period the HEPA unit will be operated without the internal filter in place (i.e., "placebo filtration"), thus blinding participants to the filters' status. The order of filtration or non-filtration will be random. At the end of each 7-day period microvascular function will be assessed, blood will be collected for assessment of systemic inflammatory markers, and urine will be collected for assessment of oxidative stress markers.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older
* Non-smoking household
* Lives in study region (Smithers or Telkwa British Columbia)

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Reactive hyperemia index | After 1 week of air filtration

SECONDARY OUTCOMES:
C-reactive protein | After 1 week of filtration

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Allen, PhD, Principal Investigator — Simon Fraser University
Locations (1):
- Simon Fraser University, Burnaby, British Columbia, Canada

REFERENCES:
- [Derived] Allen RW, Carlsten C, Karlen B, Leckie S, van Eeden S, Vedal S, Wong I, Brauer M. An air filter intervention study of endothelial function among healthy adults in a woodsmoke-impacted community. Am J Respir Crit Care Med. 2011 May 1;183(9):1222-30. doi: 10.1164/rccm.201010-1572OC. Epub 2011 Jan 21. PMID 21257787